CLINICAL TRIAL: NCT07277452
Title: Randomized Double-blind, Placebo-controlled, Multicenter Clinical Study of Nimotuzumab Combined With Nab-paclitaxel/Gemcitabine in the Perioperative Treatment of High-risk Resectable/Borderline Resectable Pancreatic Cancer
Brief Title: Nimotuzumab Combined With Nab-paclitaxel/Gemcitabine in the Perioperative Treatment of High-risk Resectable/Borderline Resectable Pancreatic Cancer
Acronym: NOTABLE-309
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IST-Nim-PC-3; NCT06781086 (obsolete NCT alias)
Record Dates: First submitted 2025-11-30; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Pancreatic Cancer, Adult
Keywords: Nimotuzumab; resectable pancreatic cancer; borderline resectable pancreatic cancer
MeSH Terms: conditions — Pancreatic cancer, adult | interventions — nimotuzumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nimotuzumab+ AG (Experimental)
  Interventions: Drug: Nimotuzumab; Drug: AG regimen
- Placebo+ AG (Placebo Comparator)
  Interventions: Drug: AG regimen; Drug: Placebo

INTERVENTIONS:
Drug: Nimotuzumab — Patients will receive 3 cycles of neoadjuvant treatment with Nimotuzumab (400 mg on days 1, 8, and 15 of a 21-day cycle), followed by surgery and 5 cycles of adjuvant Nimotuzumab (400 mg on days 1, 8, and 15 of a 21-day cycle).
  Arms: Nimotuzumab+ AG
Drug: AG regimen — Patients will receive 3 cycles of AG (gemcitabine 1000 mg/m^2 and nab-paclitaxel 125 mg/m^2 on days 1 and 8 of a 21-day cycle), followed by surgery and 5 cycles of adjuvant AG (gemcitabine 1000 mg/m^2 and nab-paclitaxel 125 mg/m^2 on days 1 and 8 of a 21-day cycle).
Drug: Placebo — Patients will receive 3 cycles of neoadjuvant treatment with placebo (400 mg on days 1, 8, and 15 of a 21-day cycle), followed by surgery and 5 cycles of adjuvant therapy (placebo 400 mg on days 1, 8, and 15 of a 21-day cycle).
  Arms: Placebo+ AG

SUMMARY:
This is a prospective, multicenter, randomized, double-blind, placebo-controlled study. Led by The First Affiliated Hospital with Nanjing Medical University and Peking University Cancer Hospital & Institute (as leading centers), its main purpose is to evaluate the clinical efficacy and safety of Nimotuzumab combined with nab-paclitaxel plus gemcitabine (AG) in the perioperative treatment of high-risk resectable/borderline resectable pancreatic cancer.

DETAILED DESCRIPTION:
This clinical study is designed as a prospective, multicenter, randomized, double-blind, placebo-controlled trial, led by two leading centers: The First Affiliated Hospital with Nanjing Medical University and Peking University Cancer Hospital & Institute. Its main purpose is to evaluate the clinical efficacy and safety of Nimotuzumab combined with nab-paclitaxel plus gemcitabine (AG regimen) in the perioperative treatment of high-risk resectable/borderline resectable pancreatic cancer. Approximately 156 patients will be enrolled in this study and randomly assigned in a 1:1 ratio to the experimental group (Nimotuzumab plus AG regimen) and the control group (placebo plus AG regimen). The primary endpoint is disease-free survival (DFS). Secondary endpoints include overall survival (OS), R0 resection rate, preoperative objective response rate (ORR), incidence of postoperative complications, and safety, etc.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 18-75 years old, gender unlimited;
* 2. Histologically or cytologically confirmed pancreatic ductal adenocarcinoma (PDAC);
* 3. Confirmed as resectable/borderline resectable pancreatic cancer by CT/MRI imaging (resectability assessment refers to NCCN guidelines). For resectable pancreatic cancer, at least one of the following high-risk factors must be met: 1) CA199 > 500 U/ml; 2) the maximum diameter of the primary tumor > 3.0 cm; 3) Severe weight loss (BMI < 18.5 kg/m² OR involuntary weight loss > 15% within 6 months); 4) Severe pain (Numeric Rating Scale [NRS]≥ 4); 5) Definite regional lymph node metastasis (N1 or N2) OR suspicious regional lymph node metastasis (short-axis diameter of lymph nodes ≥15 mm);
* 4. Voluntarily agree to sample collection (for KRAS gene testing and post-hoc analysis);
* 5. Adequate organ and bone marrow function, defined as follows: hemoglobin≥9.0 g/dL; absolute neutrophil count (ANC)≥1.5×10^9/L; platelets≥80×10^9/L; serum total bilirubin (TBIL)≤1.5×ULN; aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 times the upper limit of normal (ULN); serum creatinine≤1.5×ULN or estimated creatinine clearance > 60 mL/min;
* 6. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0-2;
* 7. Life expectancy of at least 3 months;
* 8. Women of childbearing age should have a negative result of serum HCG or urine pregnancy tests within 72 hours prior to randomization (Postmenopausal women who have had amenorrhea for at least 12 months are considered sterile and women known to have had tubal ligation are not required to undergo pregnancy tests) ;
* 9. Good compliance and signed informed consent.

Exclusion Criteria:

* 1. Previous treatment for pancreatic cancer.
* 2. Accompanied by other serious diseases, including but not limited to: active infections; unmanageable diabetes mellitus and uncontrolled hypertension (SBP>160mmHg or DBP>100mmHg); compensatory heart failure (NYHA grade III and IV), unstable angina or poorly controlled arrhythmias within 3 months prior to randomization; presence of uncontrolled pleural effusion, pericardial effusion, or ascites requiring drainage; severe portal hypertension; digestive tract obstruction; respiratory insufficiency and severe lung disease; central nervous system disease or mental illness;
* 3. Clinically diagnosed as local recurrence of pancreatic cancer, or there is evidence of peritoneal/other distant metastases;
* 4.History of other malignancies (except cured basal cell carcinoma of the skin and carcinoma in situ of the cervix);
* 5. Presence of bleeding or coagulation disorders;
* 6. Known allergy to prescription or any component of the prescription used in this study;
* 7. Known HIV infection, syphilis infection, or active hepatitis (hepatitis B or C);
* 8. Women who are pregnant or are breastfeeding;
* 9.Other reasons that are not suitable to participate in this study according to the researcher's judgment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2025-12-10 (Estimated); Primary Completion 2028-12-10 (Estimated); Study Completion 2029-12-10 (Estimated)

PRIMARY OUTCOMES:
disease-free survival (DFS) | Up to 24 months
  The time from the date of surgery to the disease recurrence or death, whichever is earlier.

SECONDARY OUTCOMES:
overall survival (OS) | Up to 24 months
  The time from the date of randomization to death due to any cause.
R0 resection rate | within 30 days after surgery
  Pathologic review will determine if an R0 resection has been performed. R0 resection indicates a microscopically margin-negative resection, in which no gross or microscopic tumor remains in the primary tumor bed.
Surgical Resection rate | within 30 days after surgery
  Patients who undergo surgical resection will be documented.
Objective response rate (ORR) | Up to 9 weeks during the neoadjuvant treatment
  Objective response rate (ORR), including complete response (CR) and partial response (PR). Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT/MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), at least a 30% decrease in the sum of the longest diameter of target lesions.
adverse events | Up to 30 days after last administration
  Frequency and severity of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Kuirong Jiang, MD, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University; Chunyi Hao, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (2):
- China (2):
  - Kuirong Jiang, Nanjing, Jiangsu
  - Chunyi Hao, Beijing